CLINICAL TRIAL: NCT04606992
Title: Combined Endoscopic and Laparoscopic Surgery (CELS) for Early Colon Cancer in High Risk Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REG-006-2020
Record Dates: First submitted 2020-10-08; First posted 2020-10-28 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-02

CONDITIONS: Colon Cancer Stage I
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Pilot feasibility
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CELS resection (Experimental): All patients included in the study will be in this arm
  Interventions: Procedure: CELS

INTERVENTIONS:
Procedure: CELS — CELS resection for early colon cancer is a compromised resection performed in frail patients

SUMMARY:
This is a pilot feasibility study on high risk patients due to frailty and comorbidity who have early stage colon cancer (UICC 1). We will use a novel resection technique with expected less risk of complications called the Combined Endoscopic and Laparoscopic Surgery (CELS). After the histopathologic evaluation. Patients will be placed in either low risk or high risk group. Depending on this, they will be followed for 3 years or referred to standard resection

DETAILED DESCRIPTION:
Combined Endoscopic and Laparoscopic Surgery (CELS) for early colon cancer in high risk patients

Investigator Morten Frederik Schlaikjær Hartwig

Local research group Ismael Gögenur Lasse Bremholm Hansen Mustafa Bulut Rasmus Dahlin Bojesen Jens Ravn Eriksen Susanne Eiholm Mads Klein Morten Rasmussen Bo Rud

International research group Phil Quirke Scarlet Brockmoeller

Background Colorectal cancer is the second most common cancer in Europe and the third most common cancer worldwide. The introduction of screening programs for colorectal cancer has resulted in an increased detection and incidence of early cancers (T1-T2). Early cancers are seen in 54% of the patients in the screening programs compared with 25 % of symptomatic patients.

Mortality rates following elective colorectal surgery range between 2.5-6% and increase for the elderly and frail patient regardless of T-stage. Nationwide morbidity rates are 16%, with approximately half of these patients requiring re-operation. The elderly patients have decreased 1-year survival leading to decreased cancer specific survival. Postoperative morbidity leads to decreased 3 year disease free survival and overall 5-year survival regardless of recurrence. Further, postoperative altered bowel function, chronic pain, and reduced quality of life affect many patients.

Numerous different scoring systems exist to assess patient frailty. Studies have shown that regardless which definition of frailty is used, the patients have a higher risk of developing adverse outcomes. Performance Status (PS) is a simple and easy to use scoring system to assess frailty. Data from DCCG has shown that performance status is independently associated with postoperative complications and death following surgery for colorectal cancer and that there is a "dose-response" relationship with increased performance score leading to higher 1-year mortality.

The risk for lymph node metastases is 8.6 % and 22 % for T1 and T2 colon cancer respectively and is dependent on several histopathological characteristics of the tumor. These histopathologic high-risk features include low tumor differentiation, lymphovascular invasion and high grade tumor budding. The presence of these features is independently related to increased risk of lymph node metastasis. If a T1 or T2 tumor has no high risk features, the risk of lymph node metastasis has been reported to be 1,2% and 3,8%respectively.

According to the Danish Colorectal Cancer Group (DCCG) annual report in 2017, there was 253 T1 and 325 T2 colon cancers. Out of these there were 84,3% and 82,9% N0 respectively. This indicates that the majority of patients with early colon cancer (ie. T1 and T2) have no benefit of additional oncological resection besides tumor excision.

Due to the low risk of lymph node metastases in early colon cancer, and the substantial risk of morbidity and mortality, local excision of the tumor could be an option in selected high risk patients (with subsequent bowel resection if final pathological evaluation shows presence of high-risk histopathological characteristics).

The Combined Endoscopic and Laparoscopic Surgery (CELS) is a novel hybrid procedure that enables large local excisions of the colon without segmental resection. It is used in some centers for local resections of large benign polyps not resectable by advanced endoscopic techniques alone such as Endoscopic Mucosal Resection (EMR).

CELS procedure Combined Endoscopic and Laparoscopic Surgery covers a variety of endoscopic procedures with simultaneous laparoscopic view and laparoscopic procedures with simultaneous endoscopic view. In our study we focus exclusively on laparoscopic resection guided by endoscopic view - an excision biopsy.

The main surgical advantage in this procedure is the ability to view the colon intra- and extraluminally simultaneously. The laparoscopic approach enables manipulation and mobilization of the colon, while the endoscopic view secures that the resection is complete and not overlapping the ileac valve or creating stenosis.

Compared to the traditional segmental oncological colon resection, the CELS resection is a minimally invasive procedure and assumed leading to a reduced surgical stress response. A RCT has compared CELS with right sided hemicolectomy and shown, shorter operating time, less intravenous fluid treatment, faster time to pass stool and shorter length of stay.

The CELS procedure has been evaluated both in retrospective and prospective randomized trials in patients with benign lesions not suitable for endoscopic resection, and is shown to be a safe procedure with comparable complication rates, but shorter convalescence and lower cost. The question is if the CELS procedure is a safe resection in the malignant tumor, as in the benign tumor.

The present study is designed to show if the CELS can be used for patients diagnosed with an early colon cancer and in high risk of operative morbidity and mortality after conventional resection due to comorbidity and frailty.

Aim The primary aim of this study is to assess feasibility and safety in high risk patients treated with CELS resection with early colon cancer.

Methods This is a non-randomized prospective feasibility study conducted at the Department of Surgery, Zealand University Hospital, Herlev University Hospital, Hvidovre University Hospital and Bispebjerg University Hospital.

The data will be collected and stored online at easytrial.net and physically at the Department of Surgery, Zealand University Hospital.

Statistical power analysis We plan to include 25 high risk patients with early colon cancer in the study. Based on data from DCCG concerning clinical tumor stage and comorbidity assessments, we expect 150 eligible patients a year in the described region of Denmark. The feasibility in the study requires that we include patients with different tumor locations throughout the colon. We believe that this will be obtained with 25 patients.

The study has started 1/3 2020 and is expected to end on the 28/2 2022.

Patient selection

Setting:

The patient has been referred to the surgical department after a colonoscopy has revealed a lesion in the colon not suitable for local endoscopic treatment and is either with endoscopic suspicion of being a cancer or there is a histological diagnosis. Usual staging will be performed with contrast enhanced CT scan of the thorax and abdomen. The patient will discussed at a MDT (Multidisciplinary Team) conference, prior to the first outpatient visit. The MDT will finally decide if the patient is a candidate for CELS resection. The patients that are included at Herlev, Hvidovre and Bispebjerg University Hospitals are reassessed at the MDT conference at Køge. Here it will finally be decided if the patient is suited for CELS resection.

If the patient meets the inclusion criteria, the patient is informed of the clinical trial orally and with written information by a medical assistant or consultant. The patient is booked and prepared for the procedure decided at the ambulatory visit.

The patient will afterwards be contacted by one of the principal investigators and given more detailed information. The informed consent is signed by the patient as described under "guidelines for obtaining well informed consent".

If the patient does not wish to participate, the patient is booked for the standard procedure at the regional hospital.

CELS procedure After introduction of general anesthesia, an orogastric tube and a foley catheter is placed. After introduction of the colonic endoscope, the abdomen is draped in sterile fashion. Then an umbilical camera port is inserted and additional ports are placed according to the location of the tumor. Standard antibiotic prophylaxis is administered intravenously.

The tumor is identified by the endoscopist. A 60mm. endo-GIA is inserted and the tumor is resected and placed in a bag intraabdominally and removed trough the umbilical port. The resection is evaluated intra- and extraluminally to ensure sufficiency and hemostasis.

The colonoscope is retracted with simultaneous desufflation. The additional laparoscopic ports are removed and the incisions closed while hemostasis is observed.

After the operation, the patient is referred to the surgical ward in an enhanced recovery setting. The patient is discharged following assessment by colorectal surgeon typically the same or next day.

The patient is referred to the surgical outpatient unit to receive the pathological assessment of the tumor and to inform of and schedule the further treatment or follow up.

After 30 and 90 days, the patient will be contacted by telephone by the principal investigator for a follow up interview.

Pathological assessment After the CELS resection, the tumor is sent as a malignant tumor specimen without conservation and as a whole resection to the Department of Pathology, Zealand University Hospital Roskilde. Here it is cast as a whole specimen and cut into relevant slides and these are evaluated. The procedure for the pathological preparation and assessment is already implemented in the clinics standard operating procedure. After the assessment of the tumor, the tumor is defined as "high-risk" or "low risk". This defines the further follow up and treatment of the patient. (For details see "Patient flow chart").

When we have included all 25 patients, the slides of the tumors are scanned and sent as pseudo-anonymized photos to the Department of Pathology, Leeds University for reassessment by Professor Philip Quirke and Dr. Scarlet Brockmoeller.

The pathological assessment is hereby evaluated as "consensus". The department of Pathology, Zealand University Hospital Roskilde will have the final decision in case there is not consensus.

The CELS patients with low risk histopathology will follow a watchful waiting (WW) program consisting of colonoscopy after 3 and 12 months, CT scans at 6, 12 and 36 months and blood sampling for circulating tumor cell DNA (CT-DNA) after 3, 6, 12 and 36 months. This is more intense than the follow up program for locally resected malignant polyps. After 1 year, the colonoscopy will be after every 5 years until the patient reaches 75 years.

The CELS patients with high risk histopathology will be referred to standard resection and subsequently placed in the regular control group for colonic cancer defined by DCCG.

Technical and practical experiences The surgical department at Zealand University Hospital Køge, performs CELS procedures on a regularly monthly basis on benign lesions. At the moment more than 70 CELS procedures have been performed at the department.

The department has over 2 years of experience with assessment of CELS operability in multidisciplinary team conferences.

Risks and side effects The literature concerning CELS for benign lesions show a general complications risk of approximately 5%. This covers both medical and surgical complications. The most frequent complication is pneumonia and urinary tract infections. Of the surgical complications, wound/port site infection is the most frequent. Bleeding from intestinal resection or skin incisions and stapling insufficiency leading to intraabdominal abscess formation has been reported.

The CELS procedure is regarded as a safe and low risk procedure.

Safety issues With regard to the benign lesions, the literature has reported 0-13% risk of local recurrence. No study has reported the recurrence for malignant resection with CELS technique. The safety of the oncological resection is of great importance in this study. Prior to the study an independent safety committee is formed by 2 external surgeons and 1 external pathologist. Every patient with a R1/R2 section or a severe complication (Clavian-Dindo≥3b) is evaluated in the committee with regard to discussion of terminating the study. The pathologist will review the specimen as a second opinion. The surgeons will evaluate the basis for decision of CELS resection, surgical procedure and postoperative treatment to ensure proper treatment. The evaluations are coordinated by the primary investigator.

If more than 4 patients have a R1/R2 resection, the study will automatically be terminated or if we experience more than 3 local recurrences with adenocarcinoma the study will be terminated.

Perspectives If this study proves that CELS is a safe and feasible treatment, the next study will be a randomized controlled trial to prove its efficacy in high risk patients. It could be the future treatment of patients with high risk morbidity and early colon cancer following the principles of personalized surgery.

Dissemination of the results Results will be presented at major endoscopy and surgery meetings and at national and international relevant congresses. The study results will be submitted for publication in international peer reviewed scientific journals with Morten Hartwig as the first author. All co-authors will adhere to the Vancouver rules.

Ethical aspects The study is approved by the National Committee on Health Research Ethics (Den Nationale Videnskabsetiske Komité) (SJ-795) and reported to the Data Protection Agency (Datatilsynet). The study is registered at www.clinicaltrials.gov. Research subjects will have to give informed consent, based on written and oral information before inclusion in the study. Participants will be informed about any side-effects, risks or unplanned events that might occur during the implementation of the study. The minimal risks will be outweighed by the potential implications for future patient care. The study will be carried out with respect to the mental and physical integrity of the participants.

Guidelines in obtaining informed consent from participants Well informed signed consent from the research subjects is an essential criterion for inclusion in the trial. Both written and oral information will be provided to each candidate to the study by either the chief investigator or other health care persons that are qualified in explaining the project in detail. The patient will be made aware of the possibility of a second person (e.g. caregiver, relative) to be present at the interview. The interview will take place in a private room in order to provide an uninterrupted communication. The detailed information on the project will be covered, in oral and written form, at the interview, including an easy-to-read presentation of the project with its predictable risks and side-effects, expected outcomes and benefits for the research.

The subjects will be entitled to some reflection time before giving consent (24-48 hours), taking care that the time limit stipulated will not interfere with the routine clinical investigations and treatments of the patient.

Sponsors The research project is initiated by, Ismail Gögenur, MD, DMSc. The study will be funded through local and national funds.

ELIGIBILITY:
Inclusion Criteria:

* UICC stage 1 colon cancer
* ASA score min. 3 and/or WHO PS score min. 1
* CELS eligible resection
* Biopsy show adenocarcinoma or suspicious lesion
* No preop chemo or radiotherapy
* Accept inclusion

Exclusion Criteria:

* Hereditary cancer
* Rectal cancer
* Radiation downstaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
Resection margin | 1 month
  R0, R1, R2

SECONDARY OUTCOMES:
Complication rate | 1 month
  30 day complication using clavian dindo grading

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Gögenur, MD, DMsc, Study Chair — University of Copenhagen
Locations (4):
- Denmark (4):
  - Bispebjerg University Hospital, Copenhagen
  - Herlev University Hospital, Herlev
  - Hvidovre University Hospital, Hvidovre
  - Zealand University Hospital, Køge

IPD SHARING:
Plan to Share IPD: No